CLINICAL TRIAL: NCT02400073
Title: Assessment of a New AutoSet Device Designed for Female Obstructive Sleep Apnea Patients on the Quality of Life of Users
Brief Title: AutoSet for Her Quality of Life Clinical Trial
Acronym: FEM-PAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA230315
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AutoSet for Her PAP device (Experimental): Patients in this study will use the AutoSet for Her: A new AutoSetting Positive Airway Pressure (PAP) device designed specifically to treat female OSA
  Interventions: Device: AutoSet for Her

INTERVENTIONS:
Device: AutoSet for Her — 3 months nightly usage of the AutoSet for Her device

SUMMARY:
Obstructive sleep apnea (OSA) has detrimental effects on the health and quality of life of suffers. Recent literature has shown that females may be particularly susceptible to adverse the quality of life effects, and that female obstructive sleep apnea manifests differently than male obstructive sleep apnea. A new AutoSetting Positive Airway Pressure (PAP) device has been designed specifically to treat female OSA. In this Cohort study, female patients who are newly diagnosed with OSA will be asked to complete various questionnaires relating to their quality of life. Patients will then use the AutoSet for Her for three months. At the completion of the three months the questionnaires will be repeated. Before treatment and after treatment quality of life will be compared to determine if treating female specific OSA in these patients improves quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Females aged ≥ 18 years
* Diagnostic PG/ PSG showing at least moderate OSA (AHI ≥ 15)
* Indication for PAP
* Participants willing and able to give written informed consent
* Ability to tolerate PAP therapy

Exclusion Criteria:

* Participants currently using CPAP or who have previous experience with CPAP
* Participants currently using supplemental oxygen
* Participants who are pregnant or planning to become pregnant in the next 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2019-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Campos-Rodríguez, Prof, Principal Investigator — Hospital Universitario de Valme
Locations (3):
- Germany (2):
  - Sleep and Ventilation Center, Blaubeuren Abbey, Ulm
  - Advanced Sleep Research GmbH, Berlin
- Hospital Universitario de Valme., Seville, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 122 patients (25 from Spain and 97 from Germany) were enrolled in the study
Period: Overall Study
Arm/Group | AutoSet for Her PAP Device
Started | 122
Completed | 111
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | AutoSet for Her PAP Device
Number analyzed (Participants) | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 97
  Spain | 25

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Quality of Life Using the Functional Outcomes of Sleep Questionnaire (FOSQ)
Description: The Functional Outcomes of Sleep Questionnaire (FOSQ) assesses quality of life based on self reported physical and mental health. The outcome measure is Change from Baseline FOSQ score at 3 months. The minimum score is 5 and the maximum score is 20. Higher scores represent a better outcome
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AutoSet for Her PAP Device
Number analyzed (Participants) | 111
score on a scale | 1.9 (3.3)

2. Secondary Outcome: Sleep Changes Assessed Through Polysomnography
Description: assessment of sleep quality (sleep efficacy, amounts of deep sleep, amounts of REM sleep). The outcome measure is changes in sleep from baseline at 3 months
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | AutoSet for Her PAP Device
Number analyzed (Participants) | 111
minutes
  change in sleep efficacy | 0.3 (2.1)
  change in deep sleep | 7 (3.1)
  change in REM sleep | 8.4 (0.5)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | AutoSet for Her PAP Device
All-Cause Mortality (participants affected / at risk) | 0/122
Serious Adverse Events (participants affected / at risk) | 0/122
Other Adverse Events (participants affected / at risk) | 0/122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No